CLINICAL TRIAL: NCT02539602
Title: Rigorous Evaluation of Need to Know (N2K): A Three-Year Quasi-Experimental Sex Education Program for High School Students in Texas
Brief Title: Evaluation of a Need to Know (N2K): A New Sex Education Program for High School Students
Acronym: N2K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC20040080E
Record Dates: First submitted 2015-08-27; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Teen Pregnancy
Keywords: High school; Longitudnal; Sexual initiation; Contraception; Adolescents; Pregnancy prevention; Sexual health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Need to Know (N2K) (Experimental): The intended dosage for treatment participants is 16 lessons (25 minutes each) each year of the program (8 in the fall and 8 in the spring). The program consists of 3 years (48 lessons) of curriculum intended for 9th, 10th and 11th grade students to be delivered in a group or classroom setting of up to 32 students. There are 16 lessons in each year of the curriculum. Eight lessons are intended to be taught in the fall semester and eight in the spring. Each lesson is 25 minutes long, and can be taught in any class period that allows for 25 minutes of content instruction.
  Interventions: Behavioral: The Need to Know students received the N2K curriculum as described previously
- Counterfactual (No Intervention): The counterfactual condition received no intervention.

INTERVENTIONS:
Behavioral: The Need to Know students received the N2K curriculum as described previously
  Arms: Need to Know (N2K)

SUMMARY:
This trial evaluated the impact of N2K, a three-year quasi-experimental study to delay sexual initiation and increase condom and contraception use among high school students. The program was administered to treatment students beginning in the fall of 2012 (9th grade) and continued through the spring of 2015 (11th grade). The purpose of this study was to measure: 1) the impact of N2K on sexual initiation at the end of the three-year program and 2) the impact of N2K on condom or contraception non-use at the end of the program.

DETAILED DESCRIPTION:
Need to Know is based on a framework of positive youth development intended to delay sexual initiation and reduce the rate of teenage pregnancy. The N2K curriculum is designed to support the treatment participants throughout their high school career with consecutive dosage for three years from 9th through 11th grade. The intended dosage for treatment participants is 16 lessons (25 minutes each) each year of the program (8 in the fall and 8 in the spring). The program consists of 3 years (48 lessons) of curriculum to be delivered in a group or classroom setting of up to 32 students. There are 16 lessons in each year of the curriculum. Eight lessons are intended to be taught in the fall semester and eight in the spring. Each lesson is 25 minutes long, and can be taught in any class period that allows for 25 minutes of content instruction.

The 9th grade course is N2K: Basics and consists of lessons that encourage self-discovery and goal setting, discuss human growth and development, adolescent risk behaviors, communication, STDs, abstinence, contraceptives, teen dating violence, legal issues, responsible media use, refusal skills, and role-playing. The 10th grade N2K: Decisions consists of lessons that increase decision making skills, clarify values, promote healthy relationships and the benefits of delaying sex, and review of anatomy, contraceptives, STDs, and legal issues. It promotes the development of critical thinking skills and application of the facts to real life situations. N2K: Decisions includes an original webisode series of 11 episodes, the first of which is viewed in class, and the others can be viewed online outside of class. The webisode series adds narrative to the basic facts being presented in class. The series runs, in conjunction with the 10th grade curriculum lessons 3-8. The 11th grade N2K: Relationships reinforces basic themes taught in prior years. It emphasizes healthy relationships, healthy living, and taking responsibility for personal health as an adolescent matures into adult life. The last three lessons are a culminating activity that allows participants to express what they have learned and present it to others. About 35% of the 48 sessions focuses on abstinence, 27% highlight positive youth development (PYD), 13% discuss risky behaviors, 12% address STDs, 8% cover contraceptives, and 5% discuss anatomy and puberty in the cumulative three years of the N2K Curriculum.

A paper and pencil survey was administered in school to assess program impacts. Treatment and comparison students were surveyed at baseline (fall 2011 for comparison and fall 2012 for treatment), and for the treatment group, surveying took place before the intervention began. Surveys were administered at the end of each year of programming (end of 9th grade, end of 10th grade, and end of 11th grade), which for the treatment students was after the N2K programming was completed for the year.

ELIGIBILITY:
Inclusion Criteria:

* Students were eligible if they were in the 9th grade in the fall of the enrollment year (2011 for comparison students, and 2012 for treatment students), and not enrolled in the LifeSkills Class, which includes students that are severely developmentally challenged. Recruits were both male and female.

Exclusion Criteria:

* Students were not eligible if they were members of the LifeSkills self-contained special education group and not mainstreamed with other students. Students in the 10th grade who were repeating a 9th grade credit(s) were excluded from Treatment survey analysis.

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1616 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Delay sexual initiation - Survey question | 3 years
  At program completion, what is the impact of Need to Know (N2K), a three-year program, on sexual initiation (vaginal intercourse) among virgins at baseline?
  Sexual initiation was measured by a survey question asking: Have you ever had sexual intercourse? Yes or No
Decreases condom or contraception non-use - Survey question | 3 years
  At program completion, what is the impact of Need to Know (N2K), a three-year program, on condom or contraception non-use for the full analytic sample?
  Condom or contraception non-use was measured by asking the following two survey questions:
  A: In the past 3 months, have you had sexual intercourse without you or your partner using a condom, even once? Yes or No
  B: In the past 3 months, have you had sexual intercourse without using an effective method of birth control, even once? Yes or No
  * Condoms
  * Birth control pills
  * The shot (Depo Provera®)
  * The patch
  * The ring (NuvaRing®)
  * IUD (Mirena or Paragard® or Skyla®)
  * Implant (Implanon® or Nexplanon®)

SECONDARY OUTCOMES:
Delay sexual initiation - Survey question | 1 year
  1. After one year, what is the impact of Need to Know (N2K), a three-year program, on sexual initiation (vaginal intercourse) among virgins at baseline?
  Sexual initiation was measured by a survey question asking: Have you ever had sexual intercourse? Yes or No
Decreases condom or contraception non-use - Survey question | 1 year
  2. After one year, what is the impact of Need to Know (N2K), a three-year program, on condom or contraception non-use for the full analytic sample?
  Condom or contraception non-use was measured by asking the following two survey questions:
  A: In the past 3 months, have you had sexual intercourse without you or your partner using a condom, even once? Yes or No
  B: In the past 3 months, have you had sexual intercourse without using an effective method of birth control, even once? Yes or No
  * Condoms
  * Birth control pills
  * The shot (Depo Provera®)
  * The patch
  * The ring (NuvaRing®)
  * IUD (Mirena or Paragard® or Skyla®)
  * Implant (Implanon® or Nexplanon®)
Delay sexual initiation - Survey question | 2 years
  3. After two years, what is the impact of Need to Know (N2K), a three-year program, on sexual initiation (vaginal intercourse) among virgins at baseline?
  Sexual initiation was measured by a survey question asking: Have you ever had sexual intercourse? Yes or No
Decreases condom or contraception non-use - Survey question | 2 years
  After two years, what is the impact of Need to Know (N2K), a three-year program, on condom or contraception non-use for the full analytic sample?
  Condom or contraception non-use was measured by asking the following two survey questions:
  A: In the past 3 months, have you had sexual intercourse without you or your partner using a condom, even once? Yes or No
  B: In the past 3 months, have you had sexual intercourse without using an effective method of birth control, even once? Yes or No
  * Condoms
  * Birth control pills
  * The shot (Depo Provera®)
  * The patch
  * The ring (NuvaRing®)
  * IUD (Mirena or Paragard® or Skyla®)
  * Implant (Implanon® or Nexplanon®)